CLINICAL TRIAL: NCT03312140
Title: Examination of the Lipid Metabolism of the Liver After Choline Substitution in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phos-CF II V1.2
Record Dates: First submitted 2017-10-04; First posted 2017-10-17 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Cystic Fibrosis Liver Disease
MeSH Terms: interventions — Choline

STUDY DESIGN:
Intervention Model Description: Pilot study to evolve the effect ot the treatment by comparing data before and after the treatment within the same patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Choline Chloride (Other): Patients receive choline chloride (1g Choline) three times a day for 12.6 weeks as a food supply
  Interventions: Drug: Choline Chloride

INTERVENTIONS:
Drug: Choline Chloride

SUMMARY:
Pilot study to investigate the effect of choline chloride in cystic fibrosis patients with liver steatosis by comparing their status before and after the intervention

DETAILED DESCRIPTION:
Within this single arm pilot study patients with cystic fibrosis and liver steatosis receive choline chloride (2x0.5 gram three times a day) as a food supply for 88 days. D9-choline metabolism is measured before and after the intervention phase. Hypothesis of the study is, that supplying choline augments the secretion of phosphatidyl choline and lipoprotein (VLDL) from the liver and therefore results in a measurable reduction of the triglyceride storage of the liver.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* male
* Cystic fibrosis is verified
* pancreatic insufficiency
* Decline of plasma phosphatidylcholine and steatosis of the liver
* informed consent is given

Exclusion Criteria:

* cirrhosis of the liver
* Hyperreactivity to choline containing food
* allergic bronchopulmonary aspergillosis or other acute exacerbations of pulmonary infections
* FEV1 < 40%
* smoker
* chronic alcohol consume
* clinically relevant diseases (for example thyroid dysfunction, disturbance of lipid metabolism, renal diseases, significant left or right ventricular functional restriction) which will change the lipid metabolism of the liver
* Implants or other reasons which make magnetic resonance examinations impossible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2016-04-24 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Measurement of D9-Methyl-Choline Kinetic | 3 months
  The substitution of choline as a food supplement will augment the phosphatidylcholine and lipoprotein (VLDL) secretion of the liver into the blood and will therefore result in a reduction of the triglyceride retention in the liver

SECONDARY OUTCOMES:
Lipid storage of the liver | 3 months
  Comparison of steatosis of the liver (measured by magnetic resonance spectroscopy or sonography) before to after the choline substitution
Augmentation of creatinine concentration within the calf muscle | 3 months
  Augmentation of creatine concentration within the calf muscle due to the choline substitution measured by magnetic resonance spectroscopy
FVC | 3 months
  Comparison of FVC before to after the choline substitution
FEV1 | 3 months
  Comparison of FEV1 before to after the choline substitution
MEF25 | 3 months
  Comparison of MEF25 before to after the choline substitution
MMEF | 3 months
  Comparison of MMEF before to after the choline substitution

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Riethmüller, PD, Principal Investigator — Klinik für Kinder- und Jugendmedizin Tübingen